CLINICAL TRIAL: NCT01109303
Title: Prospective Randomized Multicentric Trial Comparing a Static Implant and a Dynamic Implant in the Surgical Treatment of Ankle Syndesmosis Rupture
Brief Title: Static Implant Versus Dynamic Implant in the Surgical Treatment on Ankle Syndesmosis Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital de l'Enfant-Jesus (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Pelet Stephane, Dr Stephane Pelet MD, PhD Orthopedic surgeon, Hopital de l'Enfant-Jesus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEJ-446
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Ankle Syndesmosis Rupture
Keywords: ankle fracture with syndesmotic ligament rupture; ankle syndesmosis rupture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TightRope System (Active Comparator): Patients are operated on using the TightRope implant by Arthrex.
  Interventions: Procedure: TightRope System- Arthrex® / Dynamic Implant
- Screw fixation implant (Active Comparator): Patients are operated on using the rigid four-cortices 3,5 mm screw fixation by Synthes.
  Interventions: Procedure: Screw fixation - Synthes® / Static Implant

INTERVENTIONS:
Procedure: TightRope System- Arthrex® / Dynamic Implant — Patients are operated on using a dynamic implant, the TightRope System by Arthrex®. The ankle is immobilized in a plaster boot for 6 weeks.
  Arms: TightRope System
Procedure: Screw fixation - Synthes® / Static Implant — Patients are operated on using a static implant, the rigid four-cortices 3,5 mm screw fixation by Synthes®. The ankle is immobilized in a plaster boot for 6 weeks.
  Arms: Screw fixation implant

SUMMARY:
Ankle fracture is frequent and its number is increasing. In Canada, surgical treatment of these lesions is advised and the options currently used all have in common a rigid fixation of the syndesmosis which results in residual stiffness and a high level of secondary surgery, mostly to remove the implant.

The purpose of the study is to compare the treatment of ankle syndesmotic rupture by a dynamic fixation to a static fixation suggesting that the dynamic fixation method will improve the Olerud-Molander functional score of more than 15 points at the 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* men or women ≥ 18 years-old;
* ankle fracture type 44-C (AO classification) with an AP, lateral and mortise X-ray views of the ankle and an AP and lateral X-ray views of the leg;
* open fractures (Gustilo I-IIIb) or closed;
* trauma-surgery delay of less than 7 days;
* consent form signed.

Exclusion Criteria:

* ankle fractures without syndesmotic lesion;
* fracture associated with neuro-vascular lesions (Gustillo IIIc);
* pathologic fracture;
* fracture in a polytraumatized patient;
* fracture of a bone in the ipsilateral leg;
* men or women > 65 years-old;
* chronic cardiac insufficiency (ejection fraction < 30%);
* lower leg chronic venous insufficiency;
* neuro-arthropathic foot (Charcot, diabetes, etc…);
* body mass index ≥ 40;
* past medical history of fracture of the same ankle;
* medical conditions too serious for a surgery;
* men or women unfit to consent;
* any other conditions that make the examinator thinks that the follow up would be problematic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Olerud-Molander score | 3 months after surgery
  The Olerud-Molander scoring scale was chosen because it adequately represents the ankle performance following surgery (trauma or elective basis). It comprises nine functional parameters which are concerned with primary complaints, the ability to perform simple tasks and the everyday life activities.

SECONDARY OUTCOMES:
Rate of secondary surgery | within one year following surgery
  To measure the rate of secondary surgery due to infection or implant removal. Every secondary surgery during the following year counts, even for the same patient.
Radiological loss of reduction | 2 weeks after surgery
  Adequate reduction of the syndesmosis is evaluated on a simple X-ray in the anteroposterior (AP) and mortise views; the "clear space" is the distance between the medial side of fibula and the incisural surface of tibia (1 cm above tibial pilon) and cannot be more than 6 mm.
  Rate of loss of reduction and the range of this loss over 6 mm will be calculated in each group.
Implant failure | one year after surgery
  Rate of implant failure (with or without a second surgery for removal) will be measured in each group.
Radiological loss of reduction | 6 weeks after surgery
  Adequate reduction of the syndesmosis is evaluated on a simple X-ray in the AP and mortise views; the "clear space" is the distance between the medial side of fibula and the incisural surface of tibia (1 cm above tibial pilon) and cannot be more than 6 mm.
  Rate of loss of reduction and the range of this loss over 6 mm will be calculated in each group.
Radiological loss of reduction | 12 weeks after surgery
  Adequate reduction of the syndesmosis is evaluated on a simple X-ray in the AP and mortise views; the "clear space" is the distance between the medial side of fibula and the incisural surface of tibia (1 cm above tibial pilon) and cannot be more than 6 mm.
  Rate of loss of reduction and the range of this loss over 6 mm will be calculated in each group.
Radiological loss of reduction | 6 months after surgery
  Adequate reduction of the syndesmosis is evaluated on a simple X-ray in the AP and mortise views; the "clear space" is the distance between the medial side of fibula and the incisural surface of tibia (1 cm above tibial pilon) and cannot be more than 6 mm.
  Rate of loss of reduction and the range of this loss over 6 mm will be calculated in each group.
Radiological loss of reduction | 12 months after surgery
  Adequate reduction of the syndesmosis is evaluated on a simple X-ray in the AP and mortise views; the "clear space" is the distance between the medial side of fibula and the incisural surface of tibia (1 cm above tibial pilon) and cannot be more than 6 mm.
  Rate of loss of reduction and the range of this loss over 6 mm will be calculated in each group.
American Orthopaedic Foot and Ankle Society (AOFAS) score of hindfoot | 12 weeks after surgery
  An evaluation of the function (7 criteria), alignment (1 criteria) and pain (1 criteria), for a maximum of 100 points on the AOFAS scale.
AOFAS score of hindfoot | 6 months after surgery
  An evaluation of the function (7 criteria), alignment (1 criteria) and pain (1 criteria), for a maximum of 100 points on the AOFAS scale.
AOFAS score of hindfoot | 12 months after surgery
  An evaluation of the function (7 criteria), alignment (1 criteria) and pain (1 criteria), for a maximum of 100 points on the AOFAS scale.
Return to professional activities | 3 months after surgery
  This measure will be determined in days after surgery, for rate of 50% and 100% of the usual work load.
Pain on visual analog scale (VAS) | 12 weeks after surgery
  Pain is described with the VAS, which ranges from 1 to 10.
Pain on VAS | 12 weeks after surgery
  Pain is described with the VAS, which ranges from 1 to 10.
Pain on VAS | 12 months after surgery
  Pain is described with the VAS, which ranges from 1 to 10.
Range of motion | 12 weeks after surgery
  With a goniometer, a measure of the dorsal flexion (normal value 20°) and plantar flexion (40°) will be taken. Inversion and eversion will be measured according to this scale: + = weak ; ++ = middle ; +++ = complete.
Range of motion | 6 months after surgery
  With a goniometer, a measure of the dorsal flexion (normal value 20°) and plantar flexion (40°) will be taken. Inversion and eversion will be measured according to this scale: + = weak ; ++ = middle ; +++ = complete.
Range of motion | 12 months after surgery
  With a goniometer, a measure of the dorsal flexion (normal value 20°) and plantar flexion (40°) will be taken. Inversion and eversion will be measured according to this scale: + = weak ; ++ = middle ; +++ = complete.
Muscular trophicity measure of the leg | 12 weeks after surgery
  This measure is taken with a metric band 15 cm under the inferior patellar pole and must be compared to normal side. It is defined in cm with a precision of 0.5 cm. A ratio injured side/normal side will be calculated.
Muscular trophicity measure of the leg | 6 months after surgery
  This measure is taken with a metric band 15 cm under the inferior patellar pole and must be compared to normal side. It is defined in cm with a precision of 0.5 cm. A ratio injured side/normal side will be calculated.
Muscular trophicity measure of the leg | 12 months after surgery
  This measure is taken with a metric band 15 cm under the inferior patellar pole and must be compared to normal side. It is defined in cm with a precision of 0.5 cm. A ratio injured side/normal side will be calculated.
Ankle circumference measure | 12 weeks after surgery
  This measure is taken with a metric band at the bimalleolar level and must be compared to normal side. It is defined in cm with a precision of 0.5 cm. A ratio injured side/normal side will be calculated.
Ankle circumference measure | 6 months after surgery
  This measure is taken with a metric band at the bimalleolar level and must be compared to normal side. It is defined in cm with a precision of 0.5 cm. A ratio injured side/normal side will be calculated.
Ankle circumference measure | 12 months after surgery
  This measure is taken with a metric band at the bimalleolar level and must be compared to normal side. It is defined in cm with a precision of 0.5 cm. A ratio injured side/normal side will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Pelet, MD, PhD, Principal Investigator — Hôpital Enfant-Jésus
Locations (1):
- CHA-Pavillon Enfant-Jésus, Québec, Quebec, Canada